CLINICAL TRIAL: NCT00572793
Title: A Nested Case-Controlled Study Evaluating the Utility of Placental Protein 13 (PP13) In-vitro Diagnostic Kit as a Diagnostic Aiding Tool in Assessment of the Risk for Developing Preeclampsia Necessitating Delivery Before 37 Weeks (Early-preeclampsia) Based on First Trimester Blood Testing of Pregnant Women With Low and Unknown Risk
Brief Title: A Study to Evaluate the Use of Placenta Protein 13 (PP13) in the First Trimester of Pregnancy as a Diagnostic Aiding Tool in the Assessment of the Risk for Developing Preeclampsia in Women With Low and Unknown Risk
Status: Completed | Type: Observational
Sponsor: Carl Weiner, MD (Other)
Collaborators: Diagnostic Technologies Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Carl Weiner, MD, Professor and Chair, Obstetrics and Gynecology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 11063
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal serum - placental protein 13 level
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether it is possible to detect changes in the concentration of PP13 in the blood of pregnant women who may go on to develop the complication of preeclampsia later on in the pregnancy, and if these changes can be detected early enough to allow early diagnosis and treatment for prevention of these complications and reduce their damage. This study will test if the PP13 biomarker during the first trimester of pregnancy has the ability to provide assessment of risk for the development of preeclampsia that necessitates delivery before 37 weeks gestation or can predict preeclampsia before 34 weeks gestation.

DETAILED DESCRIPTION:
After obtaining informed consent maternal demographics, vital signs, height, weight, medical history, pregnancy dating, dipstick for urine protein, previous lab results, nuchal translucency results and uterine artery Doppler results (if done) will be obtained. Blood for PP13 will be obtained at 7-13 weeks and optionally at 21-23 weeks. Hospitalization and delivery information will be obtained via a chart review for evidence of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, pregnant females
* Singleton fetus at 7 0/7 to 13 6/7 weeks gestation

Exclusion Criteria:

* Multi-fetal pregnancy
* Mental retardation
* Known fetal anomaly or demise
* BMI > 35, serious medical condition

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant patients seen or referred to the obstetrical clinic
Sampling Method: Non-Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2007-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Preeclampsia necessitating delivery at gestational age < 37 weeks including HELLP syndrome and eclampsia | 37 Weeks

SECONDARY OUTCOMES:
Maternal and Neonatal morbidity and mortality and very early preeclampsia necessitating delivery before 34 weeks | 34 Weeks, At Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Carl Weiner, MD, MBA, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States